CLINICAL TRIAL: NCT03128112
Title: Using a Poster Depicting Healthy Weight to Improve Perception of Weight, a Multi-site Study
Brief Title: Healthy Weight Poster, Multi-site Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Duke University (Other); Eastgate Public Health Center (Unknown); UAB Huntsville Pediatrics (Unknown); Pediatric Associates of Northern Kentucky (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00042929
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-01

CONDITIONS: Childhood Obesity
Keywords: Parental perception, obesity, overweight
MeSH Terms: conditions — Pediatric Obesity; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exam room without poster (No Intervention): All parents will be asked to fill out a questionnaire detailing basic demographic information as well as their perception of their child's weight. Parents who are in exam rooms without posters will be ask to fill out a second short questionnaire after seeing their physician that will ask parents whether they discussed their child's weight status with their physician and whether they believe their own child is: very overweight, overweight, healthy weight, underweight, or very underweight.
- Exam room with poster (Active Comparator): All parents will be asked to fill out a questionnaire detailing basic demographic information as well as their perception of their child's weight. Parents who are in exam rooms with posters will be directed to read the poster on the exam room wall. After viewing the poster and after seeing their physician, parents will be ask to fill out a second short questionnaire that will ask parents whether they discussed their child's weight status with their physician, whether this conversation was prompted by the poster, and whether they believe their own child is very overweight, overweight, healthy weight, underweight, or very underweight.
  Interventions: Other: Exam room with poster

INTERVENTIONS:
Other: Exam room with poster — This intervention will assess whether a novel educational exam room poster can effectively prompt patients to ask pediatricians about their children's weight status and improve patents' perceptions of their children's weight status.
  Arms: Exam room with poster

SUMMARY:
This is a multi-site, cross-sectional study of 3-8 year old children and their parents presenting for a well-child check. The investigators are assessing whether a novel, educational, exam room poster can effectively prompt parents to ask their pediatricians about their children's weight status and improve parents' perceptions of their children's weight status.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether a novel, educational, exam room poster can effectively prompt parents to ask their pediatricians about their children's weight status. Exam rooms within clinics will be randomized to either have the poster or not and parents will complete questionnaires assessing weight perception, whether they discussed their child's weight with their physician, and basic demographics. Participants who are in exam rooms with a poster will also answer questions specifically about the poster.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-8 years old presenting to pediatric clinic for a well-child visit.
* Parents of include children who speak English or Spanish and are able to complete a written survey.

Exclusion Criteria:

* Parents that are <18 years old
* Children with no documented weight or height for their visit
* Any medical condition that would affect weight gain or growth such as failure to thrive, congenital heart defect, etc.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 965 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Poster assessment prompts by questionnaire | End of study - 1 year
  Assess whether the poster prompts parents to ask their child's doctor whether their child is a healthy weight.
Parents' perceptions by questionnaire | End of study - 1 year
  Assess whether the poster improves accuracy of parents' perceptions of their children's weight status.
Changes in parental perception by questionnaire | End of study - 1 year
  Among parents who view the poster, the investigators will assess whether parental perception changes differentially based on parental race/ethnicity, education, or socioeconomic background.

CONTACTS AND LOCATIONS:
Overall Officials: Callie L Brown, MD MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - UAB Health Center Huntsville, Huntsville, Alabama
  - Pediatric Associates of Northern Kentucky, Crestview Hills, Kentucky
  - Duke Children's Primary Care Brier Creek, Durham, North Carolina
  - Duke Health Center at Roxboro Street, Durham, North Carolina
  - Downtown Health Plaza, Winston-Salem, North Carolina
  - Ford Simpson Lively and Rice Pediatrics, Winston-Salem, North Carolina
  - Public Health Center - Eastgate, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doolen J, Alpert PT, Miller SK. Parental disconnect between perceived and actual weight status of children: a metasynthesis of the current research. J Am Acad Nurse Pract. 2009 Mar;21(3):160-6. doi: 10.1111/j.1745-7599.2008.00382.x. PMID 19302692
- [Background] Lundahl A, Kidwell KM, Nelson TD. Parental underestimates of child weight: a meta-analysis. Pediatrics. 2014 Mar;133(3):e689-703. doi: 10.1542/peds.2013-2690. Epub 2014 Feb 2. PMID 24488736
- [Background] Rietmeijer-Mentink M, Paulis WD, van Middelkoop M, Bindels PJ, van der Wouden JC. Difference between parental perception and actual weight status of children: a systematic review. Matern Child Nutr. 2013 Jan;9(1):3-22. doi: 10.1111/j.1740-8709.2012.00462.x. Epub 2012 Oct 1. PMID 23020552
- [Background] Moore LC, Harris CV, Bradlyn AS. Exploring the relationship between parental concern and the management of childhood obesity. Matern Child Health J. 2012 May;16(4):902-8. doi: 10.1007/s10995-011-0813-x. PMID 21594667
- [Background] Soto C, White JH. School Health Initiatives and Childhood Obesity: BMI screening and reporting. Policy Polit Nurs Pract. 2010 May;11(2):108-14. doi: 10.1177/1527154410374218. Epub 2010 Aug 2. PMID 20679328
- [Background] Wake M, Salmon L, Waters E, Wright M, Hesketh K. Parent-reported health status of overweight and obese Australian primary school children: a cross-sectional population survey. Int J Obes Relat Metab Disord. 2002 May;26(5):717-24. doi: 10.1038/sj.ijo.0801974. PMID 12032758
- [Background] Perrin EM, Jacobson Vann JC, Benjamin JT, Skinner AC, Wegner S, Ammerman AS. Use of a pediatrician toolkit to address parental perception of children's weight status, nutrition, and activity behaviors. Acad Pediatr. 2010 Jul-Aug;10(4):274-81. doi: 10.1016/j.acap.2010.03.006. Epub 2010 May 31. PMID 20554259
- [Background] Cates JR, Diehl SJ, Crandell JL, Coyne-Beasley T. Intervention effects from a social marketing campaign to promote HPV vaccination in preteen boys. Vaccine. 2014 Jul 16;32(33):4171-8. doi: 10.1016/j.vaccine.2014.05.044. Epub 2014 Jun 2. PMID 24886960
- [Background] Gee S, Chin D, Ackerson L, Woo D, Howell A. Prevalence of childhood and adolescent overweight and obesity from 2003 to 2010 in an integrated health care delivery system. J Obes. 2013;2013:417907. doi: 10.1155/2013/417907. Epub 2013 Jul 18. PMID 23970960
- [Background] Herrera J, Lockner D, Kibbe D, Marley SC, Trowbridge F, Bailey A. Innovative tools help counselors discuss childhood obesity with parents. Child Obes. 2013 Apr;9(2):144-9. doi: 10.1089/chi.2012.0095. Epub 2013 Mar 15. PMID 23496294
- [Background] Parry LL, Netuveli G, Parry J, Saxena S. A systematic review of parental perception of overweight status in children. J Ambul Care Manage. 2008 Jul-Sep;31(3):253-68. doi: 10.1097/01.JAC.0000324671.29272.04. PMID 18574384
- [Background] Towns N, D'Auria J. Parental perceptions of their child's overweight: an integrative review of the literature. J Pediatr Nurs. 2009 Apr;24(2):115-30. doi: 10.1016/j.pedn.2008.02.032. Epub 2008 Sep 5. PMID 19268233